CLINICAL TRIAL: NCT01514929
Title: A Randomized, Double-Blind, Placebo and Positive-Controlled, Crossover Study to Evaluate the Effect of IV ACHN-490 Injection on the QT/QTc Interval in Healthy Volunteers
Brief Title: A Study to Evaluate the Effect of IV ACHN-490 Injection on the QT/QTc Interval in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achaogen, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ACHN-490-006
Record Dates: First submitted 2011-11-28; First posted 2012-01-23 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Cardiac Effects in Normal Healthy Volunteers
Keywords: Thorough QT
MeSH Terms: interventions — plazomicin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Supratherapeutic Dose (Experimental): 20mg/kg ACHN-490 Injection
  Interventions: Drug: ACHN-490 Injection
- Possible Therapeutic Dose (Experimental): 15mg/kg ACHN-490 Injection
  Interventions: Drug: ACHN-490 Injection
- Moxifloxacin (Active Comparator): 400mg moxifloxacin
  Interventions: Drug: Moxifloxacin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACHN-490 Injection — 20mg/kg IV 30 minute infusion given once
  Arms: Supratherapeutic Dose
Drug: ACHN-490 Injection — 15mg/kg IV 30 minute infusion given once
  Arms: Possible Therapeutic Dose
Drug: Moxifloxacin — 400mg oral pill given once
  Arms: Moxifloxacin
Drug: Placebo — Placebo oral pill given once
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the study drug, ACHN-490 Injection, affects the QT interval in normal volunteers. The hypothesis is that the drug will not cause an increase in the QT interval.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 18 and 50 years of age and with a body mass index ≥ 18 to ≤ 33 kg/m2, and weight of ≥ 40 to ≤ 100 kg inclusive.
2. Subject is in good health as judged by the investigator based on the laboratory criteria and no clinically significant findings on the medical history or physical examination.
3. Females of child-bearing potential (defined as less than one year post-menopause) are eligible for enrollment if they are not breast feeding, they have a negative serum pregnancy test before study entry, and they are using a highly effective method of contraception for at least 3 months before study drug administration, during the study, and for at least 6 months after study completion.
4. Subjects who are willing to comply with all study activities and procedures and have provided written informed consent prior to any study procedures and have signed and dated a Health Insurance Portability and Accountability Act (HIPAA) authorization form.

Exclusion Criteria:

1. A history of additional risk factors for TdP.
2. Unstable cardiovascular disease, including recent myocardial infarction or cardiac arrhythmia.
3. Sustained supine systolic blood pressure >150 mmHg, or <110 mmHg in Part 1 or <100mmHg in Part 2, or a diastolic blood pressure >95 mmHg at screening or baseline.
4. A resting pulse rate at rest, taken during screening, of <40 bpm or >100 bpm.
5. An abnormal screening ECG indicating a second- or third-degree atrioventricular (AV) block, or one or more of the following: QRS >110 milliseconds (msec), QTcB >470 msec for females or 450 msec for males, PR interval >240 msec, or any rhythm other than sinus rhythm, which is interpreted by the Investigator to be clinically significant.
6. Uncontrolled hypertension, asthma, unstable diabetes (type I or type II), thyroid disease, seizures, myasthenia gravis, or any other neuromuscular disorder.
7. Positive results at screening for hepatitis B virus, hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infection.
8. History of central nervous system disorders, epilepsy or known seizure disorder (excluding a history of childhood febrile seizures).
9. The subject has a history of any cancer, except basal cell or stage 1 squamous cell carcinoma of the skin, which has not been in remission for at least 5 years prior to the first dose of study drug.
10. Subjects who have any condition possibly affecting drug absorption.
11. History of significant hearing loss or a family history of hearing loss, excluding age related (≥ age 65) hearing loss. A prior diagnosis of sensorineural hearing loss or Ménière's disease.
12. Clinically significant illness, including viral syndromes within 3 weeks of dosing.
13. The use of concomitant medications that prolong the QT/QTc interval.
14. Used prescription medications, over-the-counter (OTC) medications, investigational medications/therapy, vitamins, or nicotine-containing products (eg, cigarettes, cigars, chewing tobacco, snuff, etc.) within 28 days or 5 half-lives, whichever is longer, before dosing of ACHN-490 Injection.
15. Used aminoglycosides within 6 months prior to IMP administration.
16. Used herbal preparations including St. John's wort, ginseng, kava kava, ginkgo biloba, melatonin, and other nutraceuticals within 28 days prior to IMP administration.
17. Consumed caffeine- or xanthine-containing products (eg, tea, coffee, chocolate, cola, etc.), Seville oranges (sour), grapefruit, grapefruit juice, or fish liver oils within 72 hours prior to IMP administration.
18. Current participation in a clinical study of an investigational product.
19. Consumed more than 28 units of ethanol per week at any time in the 6 months before dosing (1 unit of ethanol is equivalent to 8 ounces of beer, 4 ounces of wine, or 1 ounce of spirits) or history of alcoholism and/or drug/chemical abuse. Also, consumption of any amount of ethanol within 72 hours of ACHN-490 Injection dosing.
20. Donated blood or blood components within 60 days prior to receiving study drug.
21. Women who are pregnant (or planning to become pregnant within the next 3 months) or currently breastfeeding.
22. Previous participation in this or any other ACHN-490 Injection study.
23. Known hypersensitivity to aminoglycosides or any component of the ACHN-490 Injection.
24. Subjects with poor venous access.
25. Unable to understand verbal or written English or any other language for which a certified translation of the informed consent is not available.
26. Any other medical, psychological, or social condition which, in the opinion of the PI or the medical monitor, would prevent the subject from fully participating in the study would represent a concern for study compliance or would constitute a safety concern to the subject.
27. An employee of the investigator or study center with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as a family member of the employee or investigator.
28. * (Part 1 only) * Acceptable and reproducible spirometry measurements defined as: forced expiratory volume in 1 second (FEV1) or forced vital capacity (FVC) < 80% of predicted or FEV1/FVC ratio <70% of predicted. See Appendix 7 for definitions of acceptability and reproducibility.
29. * (Part 2 only) * Known hypersensitivity to moxifloxacin or other quinolones.
30. * (Part 2 only) * Taken antacids, sucralfate, multivitamins, or other products with multivalent cations within 8 hours before oral dose in Part 2 or need to take any of the above within 4 hours after the dose administration.
31. * (Part 2 only) * Taken warfarin or Class IA or Class III antiarrhythmics within one week prior to study drug administration or expected to need to take any of the above during the study period.
32. * (Part 2 only) * Participation in Part 1 of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-10; Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety | 1 day
  In Part 1, the safety and tolerability of a single 20 mg/kg dose of ACHN-490 Injection will be assessed by measuring adverse events, blood pressure and other vital sign measurements, incidence and magnitude of clinically significant changes from baseline in clinical laboratory values (hematology, chemistry, and urinalysis), and physical examination, through 24 hours after study drug administration or resolution of all adverse events.
Effect of ACHN-490 Injection on QTcF | 24 hours
  The primary endpoint for Part 2 of this study is the time-matched change from baseline in QTcF within 24 hours of receiving study drug.

SECONDARY OUTCOMES:
PK Parameters | 24 hours
  The secondary endpoints for Part 1 of this study will include relevant PK parameters such as AUC0-t, AUC0-∞, CLT, Vss, Cmax, Tmax, and t1/2 measured for 24 hours after receiving study drug.
ECG Parameters | 24 hours
  Part 2 of the study will measure the effect of ACHN-490 Injection compared to placebo within 24 hours of study drug administration on heart rate, PR interval, QRS interval, QTcB, uncorrected QT interval, RR intervals, change in ST and T-wave morphology, and categorical change in QTc variables.
PK Parameters | 24 hours
  Part 2 of this study will measure multiple PK parameters such as AUC0-t, AUC0-∞, CLT, Vss, Cmax, Tmax, and t1/2 measured for 24 hours after receiving study drug.
Correlation between drug concentration and QTc | 24 hours
  Part 2 of this study will measure the correlation between the QTc change from baseline and plasma concentrations of ACHN-490 Injection within 24 hours of study drug administration.
Safety and tolerability | Up to 44 days
  Part 2 of this study will measure safety and tolerability of ACHN-490 Injection including adverse events, incidence and magnitude of clinically significant changes from baseline in clinical laboratory values (hematology, chemistry, and urinalysis) and physical examination; all for up to 44 days after receiving study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Achaogen, Inc.
Locations (1):
- Investigational Site, West Bend, Wisconsin, United States

REFERENCES:
- [Derived] Gall J, Choi T, Riddle V, Van Wart S, Gibbons JA, Seroogy J. A Phase 1 Study of Intravenous Plazomicin in Healthy Adults to Assess Potential Effects on the QT/QTc Interval, Safety, and Pharmacokinetics. Clin Pharmacol Drug Dev. 2019 Nov;8(8):1032-1041. doi: 10.1002/cpdd.653. Epub 2019 Jan 16. PMID 30650259